CLINICAL TRIAL: NCT06168903
Title: External Oblique Intercostal Block Versus Erector Spinae Plane Block in Laparoscopic Bariatric Surgery: A Randomized Controlled Trial
Brief Title: EOI Block Versus ESP Block in Laparoscopic Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nagy Malak , MD, Lecturer of anesthesia ,SICU and pain, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-402-2023
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Bariatric Surgery Candidate; Regional Anesthesia Morbidity
Keywords: External oblique intercostal; Erector spinae Block; Bariatric; laparoscopy

STUDY DESIGN:
Intervention Model Description: Obese patients with a body mass index (BMI) of ≥ 35 kg/m2 with comorbidities or > 40 kg/m2 and American Society of Anesthesiologists (ASA) physical status I-III and aged between 18 and 70 years scheduled for laparoscopic bariatric surgery
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be achieved using a computer-generated sequence. Concealment will be achieved using opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOI block Group (n=25):bilateral US-guided external oblique intercostal block. (Experimental): Patient in a supine position. A linear ultrasound probe will be placed in paramedian sagittal orientation between the midclavicular and anterior axillary lines at the level of the sixth rib, visualizing the external oblique and intercostal muscles. Local anesthetics are injected under the external oblique muscle.
  A 22-gauge needle will be advanced in the superomedial-to-inferolateral direction into the fascial plane between the external oblique and intercostal muscles at the caudal end of the sixth rib and between the sixth and seventh ribs.The location of the needle tip will be confirmed by hydrodissection of inter-fascial planes with 3 ml of normal saline. After negative aspiration, a total of 20 mL of bupivacaine 0.25% will be injected in the fascial plane incrementally, aspirating every 5 ml, and the block will be repeated on the other side.
  Interventions: Procedure: Ultrasound guided EOI block
- ESPB Group (n=25): bilateral US-guided erector spinae plane block (Active Comparator): Patient in a lateral position. A curvilinear ultrasound probe (5-7 MHz) will be placed transversely to identify tip of T9 transverse process 2.5-3 cm from the midline, then it will be rotated longitudinally to get a parasagittal view, visualizing the transverse process as a hyperechoic curvilinear structure with prominent finger-like acoustic shadowing beneath , lamina , spinous process, and costochondral junction medially and laterally. The erector spinae muscles are identified superficially to the tip of the T9 transverse process.The location of the needle tip will be confirmed by hydrodissection of the erector spinae muscle from the tip of the transverse process. After negative aspiration, a total of 20 mL bupivacaine 0.25% will be injected under the fascial plane incrementally, aspirating every 5 ml and the block will be repeated on the other side
  Interventions: Procedure: Ultrasound guided EOI block

INTERVENTIONS:
Procedure: Ultrasound guided EOI block — Before receiving general anesthesia, patients will be randomly assigned to one of the two study groups: the EOI block group or the ESPB group.
  Using Ultrasound (Siemens ACUSON X300 Ultrasound System), guided blocks will be administered immediately after the induction of anesthesia and prior to surgical incision by consultant anesthesiologists who have experience in regional anesthesia and are familiar with the EOI and ESPB blocks
  Other Names: Ultrasound-guided ESPB block

SUMMARY:
This study aims to compare a single shot of bilateral ultrasound-guided EOI block and ESPB in terms of intraoperative opioid consumption, postoperative pain control in the first 24 hours, and the need for rescue analgesics.

DETAILED DESCRIPTION:
The study is randomized, controlled, double blinded trial and conducted in Cairo university hospital after approval of departmental and institutional research ethics committee. Written informed consent will be obtained from all participants. Randomization will be achieved using a computer-generated sequence. Concealment will be achieved using opaque envelopes.

On arrival of the patients to operating room, patients will be secured with 20 gauge intravenous cannula. Monitoring will include ECG, non-invasive arterial blood pressure (NIBP), and pulse oximetry (SpO2). Before receiving general anesthesia, patients will be randomly assigned into one of the two study groups; EOI block Group and ESPB Group.

Induction of general anesthesia will be induced with patients in ramped position and after adequate preoxygenation using 1 µg/kg fentanyl (based on lean body weight), 2 mg/kg propofol (based on total body weight), and 0.5 mg/kg atracurium (based on the ideal body weight), in addition to 8mg IV dexamethasone for prevention of postoperative nausea & vomiting. Endotracheal intubation will be established. Anesthesia will be maintained by 1.2% MAC of isoflurane with oxygen (50%) in air and 0.1 mg/kg of atracurium will be administered every 20 minutes as maintenance anesthetic drugs. Volume-controlled ventilation will be maintained with a tidal volume of 6 mL/kg of ideal body weight and the respiratory rate will be adapted to maintain ET CO2 between 30 and 40 mmHg, and a 10 cmH2O positive end-expiratory pressure (PEEP) will be applied in all patients. Monitoring through ECG, NIBP, pulse oximetry and capnography (ETCO2) continued throughout the surgeries.

US (Siemens ACUSON X300 Ultrasound System) guided blocks will be administered immediately after the induction of anesthesia and prior to surgical incision by consultant anesthesiologists who had experience in regional anesthesia and were familiar with the EOI and ESPB blocks.

EOI block Group (n=25): this group will receive bilateral ultrasound-guided external oblique intercostal block.

The technique of ultrasound-guided EOI block will be performed with the patient in supine position. A linear ultrasound probe (4-12MHz) will be placed paramedian sagittal orientation between the midclavicular and anterior axillary lines at the level of sixth rib, visualizing the external oblique and intercostal muscles. Local anesthetics inject the under the external oblique muscle.

A 22-gauge needle will be advanced in-plane superomedial-to-inferolateral direction, into the fascial plane between the external oblique and intercostal muscles at the caudal end of the sixth rib and between the sixth and seventh ribs. The location of the needle tip will be confirmed by hydrodissection of inter-fascial planes by 3 ml of normal saline. After negative aspiration, a total of 20 mL bupivacaine 0.25% will be injected in the fascial plane incrementally, aspirating every 5 ml and the block will be repeated on the other side.

ESPB Group (n=25): this group will receive bilateral ultrasound-guided erector spinae plane block The technique of ultrasound-guided ESPB will be performed with the patient in lateral position. A curvilinear ultrasound probe (5-7 MHz) will be placed transversely to identify tip of T9 transverse process 2.5-3 cm from midline then it will be rotated longitudinally to get a parasagittal view visualizing the transverse process as a hyperechoic curvilinear structure with prominent finger-like acoustic shadowing beneath (the trident sign), with lamina (sawtooth pattern), spinous process, and costochondral junction medially and laterally. The erector spinae muscles are identified superficial to the tip of the T9 transverse process. A 22-gauge needle will be advanced in-plane craniocaudally into the fascial plane deep to erector spinae muscle. The location of the needle tip will be confirmed by hydrodissection of erector spinae muscle from tip of transverse process by 3 ml of normal saline. After negative aspiration, a total of 20 mL bupivacaine 0.25% will be injected under the fascial plane incrementally, aspirating every 5 ml and the block will be repeated on the other side.

To achieve double blinding, patients will receive the block with 40 mL bupivacaine (0.25%) by the anesthetist. Another doctor not involved in the block procedure will evaluate the patients intraoperative and postoperative.

Intraoperative inadequate analgesia, indicated by increase of HR or MAP more than 20% above preinduction baseline values, will be managed using incremental 50 microgram doses of fentanyl. Intraoperative fentanyl consumption will be calculated. All patients will receive 10 minutes before the end of surgery 1 mg granisetron or 4 mg ondansetron IV for antiemetic prophylaxis and ketorolac 30mg IV and paracetamol 1g for postoperative analgesia. At the end of surgery, muscle relaxant will be reversed using neostigmine 0.05 mg/kg and atropine 0.02 mg/kg. Awake extubation will be established after adequate reversal of neuromuscular block.

Patients will be transported to PACU and placed in the semi-sitting position, and oxygen will be given via a nonrebreathing facemask with a reservoir bag. Postoperative pain will be assessed using VAS (where 0 corresponds to no pain and 100 mm to the worst pain) at 2, 4, 6, 12, 18, and 24 hours postoperatively.

Postoperatively, all patients will receive 1 g paracetamol every 6 h, 30 mg ketorolac every 12 h.

IV morphine titration will be carried out at patient wake-up to achieve pain control (VAS ≤ 30mm) by an attending anesthesiologist blinded to group allocation. Patients with a VAS score of ≥ 40mm and patients who will request rescue analgesia will be treated with IV morphine in 2 mg increments every 5 minutes with no upper limit for the total administered dose and total morphine consumption will be recorded. If the patient appeared sedated (Ramsay sedation scale > 2), and/or severe morphine-related side effects are encountered including respiratory depression (Spo2 < 95% and/or respiratory rate < 12 breaths/min), allergic reaction, hypotension, or severe pruritus, morphine titration will be stopped and the patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients of any gender with a body mass index (BMI) of ≥ 35 kg/m2 with comorbidities or > 40 kg/m2 and American Society of Anesthesiologists (ASA) physical status I-III and aged between 18 and 70 years scheduled for laparoscopic bariatric surgery, that is, sleeve gastrectomy and/or Roux-en-Y gastric bypass (RYGB) surgery.

Exclusion Criteria:

* Coagulopathy, infection at the injection site, allergy to local anesthetics, severe hepatic or renal disease, severe cardiopulmonary disease (≥ ASA IV), diabetic or other neuropathies, patients receiving opioids for chronic analgesic therapy, and inability to comprehend visual analogue scale (VAS).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain score | 24 hours
  VAS Score at rest (static) and on movement (dynamic) at 2, 4, 6, 12, 18, and 24 hours postoperatively

SECONDARY OUTCOMES:
Time needed to perform the block | 30-60 Minutes
  Time needed to perform the block, starting from scanning to finishing on both sides.
Fentanyl consumption | Up to 4 hours
  Intraoperative fentanyl consumption
Total morphine requirements | 24 hours
  Total morphine requirements: 24 hours postoperatively.
First postoperative analgesic request | 24 hours
  Time for the first postoperative analgesic request
Postoperative nausea and vomiting | 24 hours
  Incidence of PONV
Complications related to the blocks | 24 hours
  Incidence of complications related to the blocks

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Hospitals. kasralainy, Cairo, Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No